CLINICAL TRIAL: NCT06181994
Title: Outcomes of Middle Meningeal Artery for Treatment of Chronic Subdural Hematoma; Middle Meningeal Artery Embolization for Chronic Subdural Hematoma (MESH)
Brief Title: Middle Meningeal Artery Embolization (MMAE) Outcomes for Chronic Subdural Hematoma (cSDH)
Acronym: MESH
Status: Recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Geisinger Clinic (Other); Heidelberg University (Other); Henri Mondor University Hospital (Other); Ospedale Policlinico San Martino (Other); Ospedale San Raffaele (Other); Lehigh Valley Hospital (Other); Mayo Clinic (Other); Medical University of South Carolina (Other); New York University (Other); Oregon Health and Science University (Other); Sisters of Mercy University Hospital (Other); Unity Health Toronto (Other); Sutter Health (Other); University of Iowa (Other); Thomas Jefferson University (Other); University Health Network, Toronto (Other); University Hospital, Bordeaux (Other); University of Alabama at Birmingham (Other); University of South Florida (Other); University of Washington (Other); Cornell University (Other); Westchester Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-15327
Record Dates: First submitted 2023-12-05; First posted 2023-12-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Subdural Hematoma
Keywords: Middle meningeal artery embolization; Endovascular Embolization
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multi-center retrospective cohort study aims to investigate the real-world outcomes of chronic subdural hematoma treated with MMAE, including clinical effectiveness, recurrence rates, and safety profile.

DETAILED DESCRIPTION:
Chronic subdural hematoma (cSDH) is a prevalent neurosurgical condition marked by the accumulation of blood in the subarachnoid space. Primarily affecting elderly individuals, cSDH is associated with significant morbidity and mortality rates. Current standard treatments for cSDH involve surgical evacuation through burr hole craniotomy or twist-drill craniotomy; however, recent research has illuminated the potential significance of the middle meningeal artery (MMA) in cSDH pathogenesis, suggesting an innovative minimally invasive treatment avenue. The investigator team is attempting to determine whether MMA embolization has demonstrated a favorable safety profile with a low incidence of treatment-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (18 yrs. of age or older)
* Endovascular embolization of middle meningeal artery using any embolization material:

PVA particles; Onyx, nBCA glue; dimethyl sulfoxide, microcoils, PVA with microcoils

Exclusion Criteria:

* Endovascular embolization of middle meningeal artery using any other embolization material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic subdural hematoma
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Reaccumulation of Hematoma | Within 1 month post MMAE
  The percentage of patients who were determined to have a reaccumulation of their hematoma will be tabulated and reported
Rescue surgical evacuation | Between 1-3 months post MMAE
  The percentage of patients who were determined to require rescue surgical evacuation of their hematoma will be tabulated and reported

SECONDARY OUTCOMES:
Reaccumulation of Hematoma | Between 1-3 months post MMAE
  The percentage of patients who were determined to have a reaccumulation of their hematoma will be tabulated and reported. Reaccumulation of the hematoma will be determined by measuring the hematoma thickness at a given time point and comparing it to the thickness measured at the previous time point.
Reaccumulation of Hematoma | Between 3-6 months post MMAE
  The percentage of patients who were determined to have a reaccumulation of their hematoma will be tabulated and reported. Reaccumulation of the hematoma will be determined by measuring the hematoma thickness at a given time point and comparing it to the thickness measured at the previous time point.
Reaccumulation of Hematoma | Between 6-12 months post MMAE
  The percentage of patients who were determined to have a reaccumulation of their hematoma will be tabulated and reported. Reaccumulation of the hematoma will be determined by measuring the hematoma thickness at a given time point and comparing it to the thickness measured at the previous time point.
Reaccumulation of Hematoma | Between 12-24 months post MMAE
  The percentage of patients who were determined to have a reaccumulation of their hematoma will be tabulated and reported. Reaccumulation of the hematoma will be determined by measuring the hematoma thickness at a given time point and comparing it to the thickness measured at the previous time point.
Clinical Outcome at Follow-up Clinical outcome at follow-up | Upon study discharge, 1-4 weeks
  Clinical outcome at follow-up will be assessed using a variant of the modified Rankin Scale (mRS) for neurologic disability. The classic mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome. Scoring will also include a 6 to identify patients who have expired.
Clinical Outcome at Follow-up Clinical outcome at follow-up | Within 1 month post MMAE
  Clinical outcome at follow-up will be assessed using a variant of the modified Rankin Scale (mRS) for neurologic disability. The classic mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome. Scoring will also include a 6 to identify patients who have expired.
Clinical Outcome at Follow-up Clinical outcome at follow-up | Between 1-3 months post MMAE
  Clinical outcome at follow-up will be assessed using a variant of the modified Rankin Scale (mRS) for neurologic disability. The classic mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome. Scoring will also include a 6 to identify patients who have expired.
Clinical Outcome at Follow-up Clinical outcome at follow-up | Between 3-6 months post MMAE
  Clinical outcome at follow-up will be assessed using a variant of the modified Rankin Scale (mRS) for neurologic disability. The classic mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome. Scoring will also include a 6 to identify patients who have expired.
Clinical Outcome at Follow-up Clinical outcome at follow-up | Between 6-12 months post MMAE
  Clinical outcome at follow-up will be assessed using a variant of the modified Rankin Scale (mRS) for neurologic disability. The classic mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome. Scoring will also include a 6 to identify patients who have expired.
Clinical Outcome at Follow-up Clinical outcome at follow-up | Between 12-24 months post MMAE
  Clinical outcome at follow-up will be assessed using a variant of the modified Rankin Scale (mRS) for neurologic disability. The classic mRS is a 6-point disability scale with possible scores ranging from 0-5. mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Higher scores are generally associated with less favorable outcomes. For this study patients with an mRS score of 0-2 will be determined to have had a "favorable" outcome to the procedure and patients with an mRS score of 3-5 will have been determined to have had an "unfavorable" outcome. Scoring will also include a 6 to identify patients who have expired.
Complications following MMAE | Following the procedure, up to 4 weeks
  Complications following MMAE will be identified and tabulated as either permanent or transient in nature
Timing of Complications | Following the procedure, up to 4 weeks
  Complications will be categorized and tabulated as having occurred perioperatively or postoperatively
Relatedness of Complications | Following the procedure, up to 4 weeks
  Complications will be assessed as to whether or not they were related to the surgical procedure
Duration of Hospital Stay | Upon study discharge, up to 24 months
  The median duration of hospital stay will be tabulated and reported
Clinical outcome at discharge | Upon study discharge, up to 24 months
  Clinical outcome at discharge will be assessed using the modified Rankin Scale (mRS) for neurologic disability. The mRS being used is a 7-point scale with possible scores ranging from 0-6. mRS measures the degree of disability or dependence in the daily activities of people who have suffered neurological disability. Scoring ranges from 0 (no residual symptoms) to 5 (severe neurologic disability). A patient who has expired (during or after discharge from hospital) is assigned a score of 6. Scores will be averaged and reported. Higher mRS scores are associated with progressively less favorable outcomes.
Disposition After Discharge | Upon study discharge, up to 24 months
  Disposition upon discharge will be categorized as either discharged to home; discharged to home with health service, discharged to rehabilitation facility, or death
Rescue surgical evacuation | Between 3-12 months post MMAE
  The percentage of patients who were determined to require rescue surgical evacuation of their hematoma will be tabulated and reported

CONTACTS AND LOCATIONS:
Overall Officials: David Altschul, MD, Principal Investigator — Montefiore Medical Center
Locations (19):
- United States (15):
  - Baptist Health South Florida, Inc., Coral Gables, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - University of Illinois Chicago, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - The University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC)/Harvard Medical School, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Geisinger Health, Danville, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UTHealth Houston, Houston, Texas
  - HCA Houston Healthcare Kingwood, Kingwood, Texas
- Austin Health, Heidelberg, Victoria, Australia
- Canada (3):
  - Unity Health Toronto, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No